CLINICAL TRIAL: NCT03325010
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Dose Optimization Study to Assess the Safety, Tolerability, and Efficacy of NBI-98854 for the Treatment of Pediatric Subjects With Tourette Syndrome
Brief Title: Safety, Tolerability, and Efficacy of NBI-98854 for the Treatment of Pediatric Subjects With Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBI-98854-TS2003
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Results first posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo (matching valbenazine) once daily for 12 weeks.
  Interventions: Drug: Placebo oral capsule
- Valbenazine (Experimental): Participants received valbenazine once daily for 12 weeks. The starting dose was 20 mg for participants <50 kg at baseline and 40 mg for participants ≥50 kg at baseline, and could be escalated in increments of 20 mg every 2 weeks to a maximum of 60 mg for subjects <50 kg and 80 mg for subjects ≥50 kg to achieve an optimal dose of valbenazine for each participant.
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine — vesicular monoamine transporter 2 (VMAT2) inhibitor
  Other Names: Ingrezza; NBI-98854
  Arms: Valbenazine
Drug: Placebo oral capsule — non-active dosage form
  Arms: Placebo

SUMMARY:
This is a Phase 2b, randomized, double-blind, placebo-controlled, dose-optimization study to evaluate the efficacy, safety, and tolerability of NBI-98854 titrated to the subject's optimal dose administered once daily (qd) for a total of 12 weeks of treatment in pediatric subjects with TS.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of Tourette Syndrome (TS)
2. Have at least moderate tic severity
3. Have TS symptoms that impair school, occupational, and/or social function
4. If using maintenance medication(s) for TS or TS spectrum diagnoses (e.g. obsessive-compulsive disorder [OCD], Attention-Deficit Hyperactivity Disorder [ADHD]), be on stable doses
5. Be in good general health
6. Adolescent subjects (12 to 17 years of age) must have a negative urine drug screen for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, opiates, or cannabinoids and a negative alcohol screen
7. Subjects of childbearing potential who do not practice total abstinence must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment and follow-up periods of the study

Exclusion Criteria:

1. Have an active, clinically significant unstable medical condition within 1 month prior to screening
2. Have a known history of long QT syndrome or cardiac arrhythmia
3. Have a known history of neuroleptic malignant syndrome
4. Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed)
5. Have an allergy, hypersensitivity, or intolerance to VMAT2 inhibitors
6. Have a blood loss ≥250 mL or donated blood within 30 days prior to screening
7. Have a known history of substance dependence, substance (drug) or alcohol abuse
8. Have a significant risk of suicidal or violent behavior
9. Have initiated Comprehensive Behavioral Intervention for Tics (CBIT) during the screening period or at baseline or plan to initiate CBIT during the study
10. Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (30):
  - Neurocrine Clinical Site, Sun City, Arizona
  - Neurocrine Clinical Site, Rogers, Arkansas
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Santa Clarita, California
  - Neurocrine Clinical Site, New Haven, Connecticut
  - Neurocrine Clinical Site, Hialeah, Florida
  - Neurocrine Clinical Site, Loxahatchee Groves, Florida
  - Neurocrine Clinical Site, Orange City, Florida
  - Neurocrine Clinical Site, Orlando, Florida
  - Neurocrine Clinical Site, Tampa, Florida
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, Naperville, Illinois
  - Neurocrine Clinical Site, Iowa City, Iowa
  - Neurocrine Clinical Site, Leawood, Kansas
  - Neurocrine Clinical Site, Boston, Massachusetts
  - Neurocrine Clinical Site, Lincoln, Nebraska
  - Neurocrine Clinical Site, Nashua, New Hampshire
  - Neurocrine Clinical Site, Mount Arlington, New Jersey
  - Neurocrine Clinical Site, Voorhees Township, New Jersey
  - Neurocrine Clinical Site, New York, New York
  - Neurocrine Clinical Site, The Bronx, New York
  - Neurocrine Clinical Site, Durham, North Carolina
  - Neurocrine Clinical Site, Memphis, Tennessee
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, Irving, Texas
  - Neurocrine Clinical Site, Everett, Washington
  - Neurocrine Clinical Site, Seattle, Washington
  - Neurocrine Clinical Site, Spokane, Washington
- Neurocrine Clinical Site, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled male and female pediatric participants, 6 to 17 years of age, with a Diagnostic and Statistical Manual of Mental Disorders, 4th or 5th Editions (DSM-IV or -V) diagnosis of Tourette Syndrome (TS) in the United States. The first and last participants were enrolled on 05 October 2017 and 19 July 2018, respectively.
Period: Overall Study
Arm/Group | Placebo | Valbenazine
Started | 64 | 63
Safety Analysis Set (The safety analysis set includes all participants who received at least one dose of study drug and have any post-baseline safety data collected.) | 62 | 59
Full Analysis Set (The full analysis set includes all randomized participants who have at least one evaluable change from baseline value for Total Tic Score reported at a visit (either scheduled or mapped early termination visit) during the treatment period.) | 61 | 58
Completed | 55 | 43
Not Completed | 9 | 20
Not completed — Adverse Event | 3 | 8
Not completed — Protocol Violation | 1 | 8
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Lack of Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set, which includes all randomized participants who have at least one evaluable change from baseline value for Total Tic Score reported at a visit (either scheduled or mapped early termination visit) during the treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Valbenazine | Total
Number analyzed (Participants) | 61 | 58 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.4 (2.6) | 12.2 (2.7) | 12.3 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 52 | 48 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 29
  Not Hispanic or Latino | 46 | 44 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 3 | 1 | 4
  Race: Black or African American | 8 | 1 | 9
  Race: White | 49 | 53 | 102
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Race: Other | 0 | 1 | 1
  Race: Multiple | 0 | 2 | 2
Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS) [Mean (Standard Deviation); unit: score on scale] — The YGTSS is designed to rate the overall severity of motor and phonic tic symptoms across a range of dimensions: number, frequency, intensity, complexity, and interference. The YGTSS was administered by the investigator (or qualified designee) using a computer-based structured clinical interview. The TTS is the sum of the 5 motor tic items and the 5 phonic (vocal) tic items and ranges from 0 to 50, with higher scores representing greater severity.
  score on scale | 31.2 (9.0) | 29.3 (8.7) | 30.3 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS)
Description: The YGTSS is designed to rate the overall severity of motor and phonic tic symptoms across a range of dimensions: number, frequency, intensity, complexity, and interference. The YGTSS was administered by the investigator (or qualified designee) using a computer-based structured clinical interview. The TTS is the sum of the 5 motor tic items and the 5 phonic (vocal) tic items and ranges from 0 to 50, with higher scores representing greater severity.
Time Frame: Baseline, Week 12
Population: Full analysis set, which includes all randomized participants who have at least one evaluable change from baseline value for TTS reported at a visit (either scheduled or mapped early termination visit) during the treatment period. Dose levels based on weight group and each individual participant's optimized dosing titration were prespecified to be combined within each arm.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Valbenazine
Number analyzed (Participants) | 61 | 58
score on a scale | -6.8 (1.0) | -8.9 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Valbenazine; Test type: Superiority; p = 0.1768, Mixed Models Analysis — Nominal p-value is considered statistically significant if less than 0.05. To control for multiplicity, comparisons were tested sequentially; Mean Difference (Net) = -2.1, 95% CI 2-sided [-5.2 to 1.0], Standard Error of Mean 1.5

2. Secondary Outcome: Change From Baseline to Week 12 in the Clinical Global Impression of Tics Severity (CGI-Tics-Severity) Score
Description: The CGI-Tics-Severity scale is used to assess overall severity on a 7-point scale. Each of the CGI-Tics-Severity response categories was assigned a numerical score as follows: 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill patient.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Valbenazine
Number analyzed (Participants) | 61 | 58
Score on scale | -0.7 (0.1) | -1.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Valbenazine; Test type: Superiority; p = 0.1095, Mixed Models Analysis — To control for multiplicity, comparisons were tested sequentially. Nominal p-value for this outcome measure would only be evaluated for statistical significance if the primary outcome measure was statistically significant; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.2

3. Secondary Outcome: Participants Who Are a Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS) Responder at Week 12
Description: A TTS responder is defined, on a per-visit basis, as a participant whose TTS value is reduced by at least 30% from baseline at the specified postbaseline visit.
Time Frame: Baseline, Week 12
Population: Full analysis set, which includes all randomized participants who have at least one evaluable change from baseline value for TTS reported at a visit (either scheduled or mapped early termination visit) during the treatment period. Dose levels based on weight group and each individual participant's optimized dosing titration were prespecified to be combined within each arm. Analyses include participants with outcome data available at the specified visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Valbenazine
Number analyzed (Participants) | 54 | 43
Participants | 21 | 18
Statistical Analysis 1: Comparison: Placebo vs Valbenazine; Test type: Superiority; p = 0.8190, Cochran-Mantel-Haenszel — To control for multiplicity, comparisons were tested sequentially. Nominal p-value for this outcome measure would only be evaluated for statistical significance if the primary and preceding secondary outcome measures were statistically significant; Stratified by baseline weight group (<50 kg, ≥50 kg); Risk Difference (RD) = 3.0

4. Secondary Outcome: Participants Who Are a Clinical Global Impression of Tourette Syndrome Improvement (CGI-TS-Improvement) Responder at Week 12
Description: The CGI-TS-Improvement scale is used to assess overall improvement since the initiation of study drug dosing on a 7-point scale. A CGI-TS-Improvement responder is defined, on a per-visit basis, as a participant whose CGI-TS-Improvement score is 1 ("Very much improved") or 2 ("Much improved") at the specified postbaseline visit.
Time Frame: Week 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Valbenazine
Number analyzed (Participants) | 54 | 43
Participants | 12 | 24
Statistical Analysis 1: Comparison: Placebo vs Valbenazine; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratified by baseline weight group (<50 kg, ≥50 kg); Risk Difference (RD) = 33.6

ADVERSE EVENTS:
Time Frame: Up to 14 Weeks
Arm/Group | Placebo | Valbenazine
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/62 | 0/59
Other Adverse Events (participants affected / at risk) | 17/62 | 32/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=62) | Valbenazine (N=59)
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=62) | Valbenazine (N=59)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 4 | 6
Fatigue (General disorders) | 5 | 6
Irritability (General disorders) | 2 | 3
Influenza (Infections and infestations) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 5 | 11
Somnolence (Nervous system disorders) | 0 | 11
Anxiety (Psychiatric disorders) | 2 | 3
Restlessness (Psychiatric disorders) | 0 | 3
Suicidal ideation (Psychiatric disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT03325010/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT03325010/SAP_001.pdf